CLINICAL TRIAL: NCT01045694
Title: Botulinum Toxin Versus Steroid Injection for Basal Joint Arthritis of the Thumb: a Randomized, Double Blind, Placebo-controlled Clinical Trial
Brief Title: Botulism Toxin Injection as a Treatment for Arthritis of the Basal Thumb Joint
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to acquire additional funding needed to continue this study.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1146517
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Arthritis Multiple Joint
Keywords: Carpometacarpal Joints; Osteoarthritis; Basal thumb joint arthritis; Trapeziometacarpal arthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Botulinum Toxins, Type A; Triamcinolone; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Botulinum Toxin Type A (Experimental): Arm investigates the efficacy of Botulinum Toxin A injection for the treatment of basal thumb joint arthritis
  Interventions: Drug: Botulinum Toxin Type A
- Steroid - Triamcinolone Acetonide (Active Comparator): Arm uses the standard of care - Steroid injection - as an active comparator to the experimental injection of Botulinum Toxin A for the treatment of basal thumb joint arthritis
  Interventions: Drug: Steroid - Triamcinolone Acetonide
- Lidocaine (Placebo Comparator): Arm uses plain lidocaine injection to serve as a baseline for evaluating the efficacy of Botulinum toxin as compared to steroid injection for the treatment of basal thumb joint arthritis.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Botulinum Toxin Type A — One-time injection of 50 units of Botulinum Toxin A suspended in 2 mL of normal saline, with approximately 1 mL injected or sufficient quantity to fill joint capsule
  Other Names: Botox Cosmetic; Botox
  Arms: Botulinum Toxin Type A
Drug: Steroid - Triamcinolone Acetonide — Single injection of 1 - 3 mL of 40mg/mL Triamcinolone acetonide solution
  Other Names: Kenalog-40
  Arms: Steroid - Triamcinolone Acetonide
Drug: Lidocaine — Single injection of 1 - 3 mL of 2% Lidocaine
  Other Names: Xylocaine
  Arms: Lidocaine

SUMMARY:
Basal arthritis of the thumb is a common condition with increased prevalence in post-menopausal women, obese persons, and the elderly. Surgical options are varied and efficacious, but not all patients are candidates for surgery. The successes and pitfalls of previous, similar trials are carefully considered in the creation of our own. Though steroid injection is the standard of care in basal joint arthritis, current data does not support its efficacy beyond placebo effect. No trial has yet examined the efficacy of botulinum toxin type A (BTX-A) injection into the basal thumb joint nor compared it to steroid. Since efficacy of steroid is questionable at best, our hope is that BTX-A injection of the basal joint might be the next great tool in treating this common, debilitating disease.

DETAILED DESCRIPTION:
Purpose: Basal joint arthritis, or carpometacarpal (CMC) osteoarthritis, of the thumb is very common, particularly in the elderly. Morbidities include pain, decreased range of motion, and decreased strength. Nonsurgical treatments for CMC arthritis include oral analgesics, splinting, and steroid injection. In multiple recent trials, botulinum toxin A (BTX-A) injection has been shown to be an efficacious nonsurgical option for osteoarthritis of large joints, including those that have failed steroid injections. To our knowledge, the efficacy of BTX-A injection in thumb CMC arthritis has not been examined.

Methods: Patients with a clinical and radiographic diagnosis of basal joint arthritis who are appropriate and willing candidates for injection therapy will be selected. The primary symptom indicating need for injection would be pain not controlled with more conservative measures (e.g. nonsteroidal anti-inflammatory drugs (NSAIDs), splinting, physical therapy, etc.) Weakness and impaired functioning are also considered. Exclusion criteria will include any injection within the last 12 months or surgical treatment. All patients will undergo Eaton staging radiographically prior to treatment. Informed consent will be obtained and patients will be randomly assigned to one of three groups. One group will receive BTX-A injections, the second group will receive triamcinolone plus lidocaine injections, and the third group will receive saline plus lidocaine injections of the thumb CMC joint. Prior to treatment, patients' baseline function will be assessed with pinch, grip, and range of motion measurements, and the affect of their disease will be measured with a visual analog pain scale and the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. Pain scales and DASH questionnaires will be completed at twenty-four hours, ten days, twelve weeks, six months, and one year after treatment. Pain scales will be recorded for average pain and maximum pain. Clinical evaluations with pinch, grip, and range of motion measurements will occur ten days, twelve weeks, six months, and one year after treatment. All patients will be asked to return when sufficient symptoms recur to warrant further treatment.

Expected Results: We hypothesize that BTX-A injection will have equal or better efficacy than steroid injection for the treatment of basal joint arthritis.

Expected Conclusion: No study to date has examined BTX-A as a treatment for basal joint arthritis. Some patients are not surgical candidates and are reliant on non-surgical treatments for pain control and maintenance of function. BTX-A has shown to be effective in treating osteoarthritis of larger joints that undergo frequent use, including cases resistant to steroid injections. The basal thumb joint also undergoes frequent use and is often resistant to steroid injection. We believe that BTX-A will provide another efficacious non-surgical option for treatment of the CMC joint of the thumb. We estimate that the study will require approximately three to four years to achieve adequate patient numbers for each group.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence of basal joint arthritis
* Associated symptoms of basal joint arthritis including:
* Pain
* Decreased range of motion
* Decreased thumb strength

Exclusion Criteria:

* Persons under the age of 18
* Women who are currently pregnant
* Incompetent persons or persons otherwise incapable of effectively communicating the subjective experience of pain
* Prior surgery on the joint
* Injection in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H. Colbert, MD, Principal Investigator — University of Missouri-Department of Surgery-Division of Plastic Surgery
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 8 enrollments: 6 completed and 2 withdrew voluntarily. Study was terminated early due to lack of funds. No data analysis was completed.
Pre-assignment Details: 8 participants were randomized; 2 withdrew voluntarily. Study was terminated due to lack of funds, and unblinding did not occur - it is not known how many participants were placed in each group.
Groups:
- Arthritis Treatment: Participants received one of three treatments:
  * Botulism Toxin Type A: One-time injection of 50 units of Botulinum Toxin A suspended in 2 mL of normal saline, with approximately 1 mL injected or sufficient quantity to fill joint capsule
  * Lidocaine: Single injection of 1 - 3 mL of 2% Lidocaine
  * Triamcinolone Acetonide: Single injection of 1 - 3 mL of 40mg/mL Triamcinolone acetonide solution
Period: Overall Study
Arm/Group | Arthritis Treatment
Started | 8
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 8 participants were randomized; 2 withdrew voluntarily. Study was terminated due to lack of funds, and unblinding did not occur - it is not known how many participants were placed in each group.
Arm/Group | Arthritis Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Pain
Time Frame: twenty-four hours, ten days, twelve weeks, six months, and one year
Population: 8 participants were randomized; 2 withdrew voluntarily. Study was terminated due to lack of funds, and unblinding did not occur - it is not known how many participants were placed in each group. Data was not collected or analyzed.
Arm/Group | Arthritis Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Range of Motion
Time Frame: twelve weeks, six months, and one year
Population: as for outcome 1
Arm/Group | Arthritis Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Strength
Time Frame: twelve weeks, six months, and one year
Population: as for outcome 1
Arm/Group | Arthritis Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Arthritis Treatment: Participants received one of three treatments:
  * Botulism Toxin Type A: One-time injection of 50 units of Botulinum Toxin A suspended in 2 mL of normal saline, with approximately 1 mL injected or sufficient quantity to fill joint capsule
  * Lidocaine: Single injection of 1 - 3 mL of 2% Lidocaine
  * Triamcinolone Acetonide: Single injection of 1 - 3 mL of 40mg/mL Triamcinolone acetonide solution
    8 participants were randomized; 2 withdrew voluntarily. Study was terminated due to lack of funds, and unblinding did not occur - it is not known how many participants were placed in each group.
Arm/Group | Arthritis Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of funds and no data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes